CLINICAL TRIAL: NCT00770796
Title: Usefulness of Atorvastatin (80 mg) in Prevention of Contrast-Induced Nephropathy in Patients With Chronic Renal Disease
Brief Title: Statins for Prevention of Contrast Induced Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ospedale Misericordia e Dolce (Other)
Responsible Party: Principal Investigator, Mauro Maioli, MD, Ospedale Misericordia e Dolce
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Prato0702
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Contrast Induced Nephropathy
Keywords: Contrast induced nephropathy
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo
- Atorvastatin (Active Comparator): 80 mg die of Atorvastatin given at least two days before elective angiography or angioplasty and continued for two days after.
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — 80 mg die
  Arms: Atorvastatin
Drug: Placebo
  Arms: Placebo

SUMMARY:
In this randomized study the investigators wish to explore the role of pre-procedural statin therapy for the prevention of contrast induced nephropathy in patients with moderate-to-severe renal dysfunction, submitted to elective coronary or angioplasty.

ELIGIBILITY:
Inclusion Criteria:

* patients with pre-angiographic estimated creatinine clearance < 60 ml/min

Exclusion Criteria:

* contrast medium administration within the previous 10 days
* end-stage renal failure requiring dialysis
* refusal to give informed consent
* previous therapy with statin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2006-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Contrast-induced nephropathy was defined as an absolute increase of at least 0.5 mg/dl from the baseline value in serum creatinine concentration within the first 24 hours after contrast exposure and peaking up to 5 days afterwards | within 5 days after contrast exposure

SECONDARY OUTCOMES:
Relative increase ≥ 25% over baseline serum creatinine within 5 days after contrast agent administration | within 5 days after contrast agent administration
Adverse clinical events within 1 month, including in-hospital death and need for dialysis or hemofiltration | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Maioli, MD, Principal Investigator — Ospedale Misericordia e Dolce, Prato